CLINICAL TRIAL: NCT06836583
Title: ULTRASOUND-GUIDED PERCUTANEOUS VERSUS TRANS-NASAL PTERYGOPALATINE FOSSA BLOCK in ENDOSCOPIC TRANS-SPHENOIDAL PITUITARY GLAND SURGERY: RANDOMIZED CONTROLLED TRIAL
Brief Title: Sphenopalatine Ganglion Block in Endoscopic Transphenoidal Pituitary Gland Surgery
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Donia Hany Saad, Lecturer of anaesthesia and surgical ICU, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sphenopalatine ganglion block
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: ULTRASOUND-GUIDED PERCUTANEOUS VERSUS TRANS-NASAL PTERYGOPALATINE FOSSA BLOCK in ENDOSCOPIC TRANS-SPHENOIDAL PITUITARY GLAND SURGERY
Keywords: sphenopalatine ganglion block; transphenoidal pituitary gland surgery; ultrasound guided sphenopalatine ganglion block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bilateral trans-nasal pterygopalatine Fossa block (Active Comparator): using 4ml 0.25% bupivacaine after the induction of GA.
  Interventions: Other: trans-nasal pterygopalatine Fossa block
- Bilateral US-guided infrazygomatic percutaneous pterygopalatine Fossa block (Active Comparator): using 4ml 0.25% bupivacaine after the induction of GA
  Interventions: Other: US-guided infrazygomatic percutaneous pterygopalatine Fossa block

INTERVENTIONS:
Other: trans-nasal pterygopalatine Fossa block — Patients will be placed in 15-degree reverse Trendelenburg position, between the middle and inferior turbinates. This passage will be sterilized by an cotton-tipped applicator soaked with iodine solution. A 20-gauge/5-inch spinal needle will be used after bending 2-3 mm of its tip along the port side with a sterile needle holder to form a 45 angle. The needle will be lubricated with 5% lidocaine jelly, inserted into the nasal meatus and advanced with the bevel pointer facing laterally. Under endoscopic control (0_ optics, 4 mm diameter), the needle will be inserted between middle and inferior turbinate. A total of 4 ml 0.25% bupivacaine will be injected after negative aspiration just behind and over middle turbinate tail, where the pterygopalatine fossa is deeply located.
  Arms: Bilateral trans-nasal pterygopalatine Fossa block
Other: US-guided infrazygomatic percutaneous pterygopalatine Fossa block — US- guided percutaneous PPFB:
  Patients will be placed in the lateral head position; the patient's mouth is slightly opened. Following standard sterile preparations, US linear probe covered with sterile sheath is positioned horizontally on the side of the face just below the zygomatic bone superior to the mandibular notch and anterior to the mandibular condyle to visualize the coronoid process, the lateral pterygoid muscle, the lateral pterygoid plate, and the maxillary bone, and the maxillary artery. Needle will be inserted in-plane parallel to the transducer probe and advanced from medial to lateral toward the pterygopalatine fossa. Following negative aspiration, the injectate is deposited deep to the lateral pterygoid muscle and plate. A total of 4 ml 0.25% bupivacaine will be injected.
  Arms: Bilateral US-guided infrazygomatic percutaneous pterygopalatine Fossa block

SUMMARY:
The primary aim of this study is to compare the effect of bilateral US guided percutaneous PPFB versus transnasal approach on intraoperative anaesthetic requirements (guided by entropy) in patients undergoing endoscopic transsphenoidal resection of pituitary gland surgery in conjucation with general anaesthesia (GA).Secondary aims: total dose of intraoperative dexmedetomidine, intraoperative analgesia (fentanyl), haemodynamics, the surgical field conditions, recovery pattern, and side effects

DETAILED DESCRIPTION:
Endoscopic endonasal transsphenoidal resection of pituitary gland is the currently most used method for the resection of pituitary tumors. It is a minimally invasive surgical technique to access sellar and parasellar lesions.

The main goal in endoscopic pituitary surgery are minimal tissue manipulation and clear bloodless field with better panoramic visualization under haemodynamic stability and good postoperative analgesia to improve the outcome .pterygopalatine fossa block (PPFB) is used to maintain haemodynamic stability and to decrease intraoperative anaesthetic requirements (PPFB)can be done transnasal or percutaneous ultrasound guided

ELIGIBILITY:
Inclusion Criteria:

* patients belonging to American Society of Anesthesiologists (ASA) class I or II
* patients scheduled for Endoscopic Transphenoidal Pituitary gland Surgery

Exclusion Criteria:

Patients will be excluded if; .History of allergy or contraindication to any of the studied drugs.

* Patients for whom pterygopalatine fossa block is contraindicated (patient refusal, fascial anomalies, coagulation disorder, skin infection at the injection site) .Obese patients with BMI more than 35 Kg/m2.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-27 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Intraoperative anaesthetic requirements (guided by entropy) in patients undergoing endoscopic transsphenoidal resection of pituitary adenoma in conjucation with general anaesthesia (GA). | recorded after 15 minutes from the induction of anaesthesia, then every 15 minutes till the end of the surgery. Total volume of anaesthetic agent will be measured at the end of the surgery (millimeter /minutes).
  The primary aim of this study is to compare the effect of bilateral US guided percutaneous PPFB versus transnasal approach on intraoperative anaesthetic requirements (guided by entropy) in patients undergoing endoscopic transsphenoidal resection of pituitary gland surgery in conjucation with general anaesthesia (GA).

IPD SHARING:
Plan to Share IPD: No